CLINICAL TRIAL: NCT04348253
Title: Reconstruction of Chronic Scapholunate Ligament Injuries in the Wrist: A Randomized Controlled Trial Comparing The Berger Capsulodesis and Three-Ligament-Tenodesis (3LT)
Brief Title: Danish Multicenter Scapholunate Ligament Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-10-72-169-18
Record Dates: First submitted 2020-03-30; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-03

CONDITIONS: Ligament Injury; Wrist Sprain

STUDY DESIGN:
Intervention Model Description: randomized trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Scares are identical. Patient and examiner are blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Berger (Active Comparator): Bergers capsulodesis
  Interventions: Procedure: Berger
- 3LT (Active Comparator): Three ligament tenodesis
  Interventions: Procedure: 3LT

INTERVENTIONS:
Procedure: Berger — Treatment 1
  Arms: Berger
Procedure: 3LT — Treatment 2
  Arms: 3LT

SUMMARY:
Comparison of two surgical techniques commonly used for reconstruction of the scapholunate (SL) ligament. A randomized multicenter study.

DETAILED DESCRIPTION:
This multicentre study aim to compare two surgical techniques commonly used for reconstruction of the scapholunate (SL) ligament. The investigators compare patient reported, clinical and radiological outcomes up to 10 years after treatment of complete dynamic or static but reducible SL ligament lesions. The participants are randomized to two treatments. Effect parameters before and after intervention are compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years (both included).
* Symptomatic SL instability (VAS score ³3, QDASH score ³ 20).
* > 6 weeks since symptomatic hand trauma (chronic SL lesions).
* SL gapping on radiographic stress views or SL gapping (³2mm) on static PA views.
* Complete SL ligament lesion confirmed by wrist arthroscopy

Exclusion Criteria:

* Geissler grade 1-3 SLL injury (evaluated by arthroscopy).
* Concomitant complete luno-triquetral (LT) ligament injury (evaluated by arthroscopy).
* Lesion of TFCC leading to DRUJ instability (evaluated by arthroscopy).
* Radiocarpal or midcarpal arthritis evaluated by arthroscopy.
* Previous fracture in carpus or intraarticular radius fracture with step off (³2 mm), disposing to posttraumatic arthritis.
* Adverse effects after extra articular radial fractures (dorsal angulation ³10 grader).
* Peroperatively non-reducible scaphoid flexion/SL gap.
* Terminal illness or severe medical illness: ASA score higher than or equal to 3.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2033-04-30 (Estimated)

PRIMARY OUTCOMES:
The Disabilities of the Arm, Shoulder and Hand Score (QuickDash) | At all follow-ups (0-10 years)
  points

SECONDARY OUTCOMES:
Grip-strength | At all follow-ups (0-10 years)
  kg
SL angle | At all follow-ups (0-10 years)
  degrees
The Patient-Rated Wrist Evaluation (PRWE) score | At all follow-ups (0-10 years)
  points
Wrist motion | At all follow-ups (0-10 years)
  degrees

CONTACTS AND LOCATIONS:
Overall Officials: Janni K Thillemann, Dr, Principal Investigator — Hospitalsenheden Vest
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Hospital Unit Vest, Holstebro

IPD SHARING:
Plan to Share IPD: No